CLINICAL TRIAL: NCT05018130
Title: Bio-Integrative Versus Metallic Screws for Calcaneus Osteotomies: A Non- Inferiority Randomized Clinical Trial
Brief Title: Bio-Integrative Versus Metallic Screws for Calcaneus Osteotomies
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, John Femino, Assistant Professor, University of Iowa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202106228
Record Dates: First submitted 2021-08-10; First posted 2021-08-24 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-08

CONDITIONS: Flatfoot; Bone Resorption; Cavus Deformity; Osteolysis; Complication
Keywords: Bone Healing; Osteotomy; Calcaneus; Bio-integrative; Metallic; Screws
MeSH Terms: conditions — Flatfoot; Bone Resorption; Talipes Cavus; Osteolysis

STUDY DESIGN:
Intervention Model Description: Randomized, investigator-blinded, in parallel groups, two-arms, single-center, non-inferiority, clinical trial.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The evaluator doctor will not have access to the protocol test applied to each patient and the surgeries will be conducted by different physicians.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bio-integrative (Experimental): Traditional oblique calcaneus osteotomy through a lateral approach. After a 10mm displacement, the osteotomy will be fixed with two 4.0mm bio-integrative cannulated screws.
  Interventions: Procedure: Calcaneus Osteotomy (Bio-integrative)
- Metallic (Active Comparator): Traditional oblique calcaneus osteotomy through a lateral approach. After a 10mm displacement, the osteotomy will be fixed with two 4.0mm metallic cannulated screws.
  Interventions: Procedure: Calcaneus Osteotomy (Metallic)

INTERVENTIONS:
Procedure: Calcaneus Osteotomy (Metallic) — Calcaneus Displacement Osteotomy using two metallic screws
  Arms: Metallic
Procedure: Calcaneus Osteotomy (Bio-integrative) — Calcaneus Displacement Osteotomy using two bio-integrative screws
  Arms: Bio-integrative

SUMMARY:
The use of bio-integrative implants in orthopedic surgery is growing exponentially. As many biomechanical and histological studies were able to sustain its structural and biological properties, few clinical studies are available to support its advantages, such as good osteosynthesis, lower rates of removal, and diminished implant-related artifact in imaging studies. This information is vital to providers when choosing the proper material and planning postoperative treatment. This trial intends to test the capacity of the bioabsorbable screws in reaching the same clinical and radiographical outcomes of the current metallic screws.

DETAILED DESCRIPTION:
A minimum of 44 patients undergoing Medial or Lateral Displacement Calcaneal Osteotomy (MDCO) will be randomized in two parallel groups for surgery, considering applied the implant. One group will be operated using two 4.0mm cannulated bio-integrative (absorbable) screws, and the other group using two 4.0mm cannulated metallic screws. Patients will be blinded evaluated for a mean follow-up of twelve weeks in terms of bone healing, complications, and implant-related artifact using weight-bearing computed tomography (WBCT).

ELIGIBILITY:
Inclusion Criteria:

* Individuals must be older than 18 and younger than 75 years of age, both genders;
* Participants must be experiencing symptoms related to their baseline condition for at least six months before the surgery;
* Clinical diagnosis of hindfoot malignment, defined as the presence of a clinical hindfoot angle above 10 degrees of valgus or any degree of varus;
* Surgical planning, including a calcaneus displacement osteotomy through a traditional oblique cut.

Exclusion Criteria:

* Previous surgery involving the affected calcaneus;
* History or documented evidence of autoimmune or peripheral vascular diseases;
* History or documented evidence of peripheral neuropathy (nervous compression syndrome, tarsal tunnel syndrome) or systemic inflammatory disease a (rheumatoid arthritis, spondylitis, Reiter Syndrome, etc.);
* Any condition that represents a contraindication of the proposed therapies;
* Impossibility or incapacity to sign the informed Consent Form;
* Presence of infectious process (superficial on the skin and cellular tissue, or deep in the bone) in the region to be treated.
* Osteotomies requiring resection of wedges (Dweyer, triple Dweyer, etc.);
* Osteotomies planned to occur in a non-traditional cut (Malerba, Scarf, etc.).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2024-07-30 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Bone healing | 6 weeks
  - Amount of bone bridging crossing the osteotomy site:
  Determined by the percentage of bone trabeculae crossing the osteotomy site on every tomography cut (amount of the cut in millimeters that shows bone spanning the two fragments divided by the total amount of osteotomy's surface on the cut).
  - Weight-bearing computed tomography (WBCT) acquisitions will be used to determine this percentage.

SECONDARY OUTCOMES:
Complications | 6 weeks
  - Percentage of minor and major complications:
  Dehiscence: inability to heal the soft tissue coverage until the end of the 4th post-operative week.
  Peripherical nerve damage: hypoesthesia or paresthesia not solved until the 6th week after the surgery.
  Infection: clinical signs of site infection or pus drainage at the wound that required antibiotics.
Implant-related artifact | 6 weeks
  - Quantity of Hounsfield units around the implants
  Measured on WBCT acquisitions.

CONTACTS AND LOCATIONS:
Overall Officials: Nacime Salomao Barbachan Mansur, Study Director — Visiting Associate
Locations (1):
- Departament of Orthopaedics and Rehabilitation, University of Iowa, Carver College of Medicine, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Yes
Nonidentified data will be shared to researchers upon request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After the study's publication and for 10 years.
Access Criteria: Reasonable request.

REFERENCES:
- [Background] Acar B, Kose O, Unal M, Turan A, Kati YA, Guler F. Comparison of magnesium versus titanium screw fixation for biplane chevron medial malleolar osteotomy in the treatment of osteochondral lesions of the talus. Eur J Orthop Surg Traumatol. 2020 Jan;30(1):163-173. doi: 10.1007/s00590-019-02524-1. Epub 2019 Aug 2. PMID 31375999
- [Background] Cicchinelli LD, Stalc J, Richter M, Miller S. Prospective, Multicenter, Clinical and Radiographic Evaluation of a Biointegrative, Fiber-Reinforced Implant for Proximal Interphalangeal Joint Arthrodesis. Foot Ankle Orthop. 2020 Nov 27;5(4):2473011420966311. doi: 10.1177/2473011420966311. eCollection 2020 Oct. PMID 35097414
- [Background] Daghino W, Bistolfi A, Aprato A, Masse A. Bioabsorbable implants in foot trauma surgery. Injury. 2019 Aug;50 Suppl 4:S47-S55. doi: 10.1016/j.injury.2019.01.016. Epub 2019 Jan 23. PMID 30711319
- [Background] Hovis WD, Bucholz RW. Polyglycolide bioabsorbable screws in the treatment of ankle fractures. Foot Ankle Int. 1997 Mar;18(3):128-31. doi: 10.1177/107110079701800303. PMID 9116891
- [Background] Park S, Kim JH, Kim IH, Lee M, Heo S, Kim H, Kim EH, Choy YB, Heo CY. Evaluation of poly(lactic-co-glycolic acid) plate and screw system for bone fixation. J Craniofac Surg. 2013 May;24(3):1021-5. doi: 10.1097/SCS.0b013e31827fee09. PMID 23714938
- [Background] Partio N, Mattila VM, Maenpaa H. Bioabsorbable vs. titanium screws for first tarsometatarsal joint arthrodesis: An in-vitro study. J Clin Orthop Trauma. 2020 May-Jun;11(3):448-452. doi: 10.1016/j.jcot.2019.08.017. Epub 2019 Aug 28. PMID 32405207
- [Background] Qi L, Chang C, Xin T, Xing PF, Tianfu Y, Gang Z, Jian L. Double fixation of displaced patella fractures using bioabsorbable cannulated lag screws and braided polyester suture tension bands. Injury. 2011 Oct;42(10):1116-20. doi: 10.1016/j.injury.2011.01.025. Epub 2011 Feb 22. PMID 21345433
- [Background] Tanner MC, Heller R, Westhauser F, Miska M, Ferbert T, Fischer C, Gantz S, Schmidmaier G, Haubruck P. Evaluation of the clinical effectiveness of bioactive glass (S53P4) in the treatment of non-unions of the tibia and femur: study protocol of a randomized controlled non-inferiority trial. Trials. 2018 May 30;19(1):299. doi: 10.1186/s13063-018-2681-9. PMID 29843766
- [Background] Zhang J, Xiao B, Wu Z. Surgical treatment of calcaneal fractures with bioabsorbable screws. Int Orthop. 2011 Apr;35(4):529-33. doi: 10.1007/s00264-010-1183-5. Epub 2011 Jan 5. PMID 21207026
- [Background] Jones CP, Coughlin MJ, Shurnas PS. Prospective CT scan evaluation of hindfoot nonunions treated with revision surgery and low-intensity ultrasound stimulation. Foot Ankle Int. 2006 Apr;27(4):229-35. doi: 10.1177/107110070602700401. PMID 16624210